CLINICAL TRIAL: NCT02847169
Title: Clinical Performance of Toric Hydrogel Contact Lenses Following One Week of Daily Wear
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: CooperVision, Inc. (Industry)
Responsible Party: Sponsor
Organization: CooperVision International Limited (CVIL) (Industry)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: EX-MKTG-66
Record Dates: First submitted 2016-07-25; First posted 2016-07-28 (Estimated); Results first posted 2017-05-08 (Actual); Last update posted 2017-05-08 (Actual); Status verified 2017-03

CONDITIONS: Astigmatism
MeSH Terms: conditions — Astigmatism

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- filcon IV1 toric lens (Active Comparator): Participants are randomized to wear filcon IV1 toric lens pair for 1 week during the cross over study.
  Interventions: Device: filcon IV1 toric lens
- ocufilcon D toric lens (Active Comparator): Participants are randomized to wear ocufilcon D toric lens pair for 1 week during the cross over study.
  Interventions: Device: ocufilcon D toric lens

INTERVENTIONS:
Device: filcon IV1 toric lens — toric contact lens
  Arms: filcon IV1 toric lens
Device: ocufilcon D toric lens — toric contact lens
  Arms: ocufilcon D toric lens

SUMMARY:
The aim of this prospective study is to evaluate the clinical performance of filcon IV1 toric and ocufilcon D toric contact lenses after 1 week of wear in each pair.

DETAILED DESCRIPTION:
This is a 30-subject, prospective, randomized, double masked, bilateral, 1 week cross-over study comparing the fitting characteristics of filcon IV1 toric lenses against ocufilcon D hydrogel toric lenses.

ELIGIBILITY:
Inclusion Criteria:

* A person is eligible for inclusion in the study if he/she:

  * Is between 18 and 40 years of age (inclusive)
  * Has had a self-reported visual exam in the last two years
  * Is an adapted soft toric contact lens wearer
  * Has a contact lens spherical prescription between +6.00 to - 9.00 (inclusive)
  * Have no less than -0.75D of astigmatism and no more than -2.00 D in both eyes.
  * Can achieve best corrected spectacle distance visual acuity of 20/25 (0.10 logMAR) or better in each eye.
  * Can achieve a distance visual acuity of 20/30 (0.18 logMAR) or better in each eye with the study contact lenses.
  * Has clear corneas and no active ocular disease
  * Has read, understood and signed the information consent letter.
  * Patient contact lens refraction should fit within the available parameters of the study lenses.
  * Is willing to comply with the wear schedule (at least 5 days per week, > 8 hours/day assuming there are no contraindications for doing so).
  * Is willing to comply with the visit schedule

Exclusion Criteria:

* A person will be excluded from the study if he/she:

  * Has a CL prescription outside the range of the available parameters of the study lenses.
  * Has a spectacle cylinder less than -0.75D or more than -2.00 D of cylinder in either eye.
  * Has a history of not achieving comfortable CL wear (5 days per week; > 8 hours/day)
  * Has contact lens best corrected distance vision worse than 20/25 (0.10 logMAR) in either eye.
  * Presence of clinically significant (grade 2-4) anterior segment abnormalities
  * Presence of ocular or systemic disease or need of medications which might interfere with contact lens wear. Confidential EX-MKTG-66 Clinical Performance of Toric Hydrogel Contact Lenses Following One Week of Daily Wear 10
  * Slit lamp findings that would contraindicate contact lens wear such as:

    * Pathological dry eye or associated findings
    * Pterygium, pinguecula, or corneal scars within the visual axis
    * Neovascularization > 0.75 mm in from of the limbus
    * Giant papillary conjunctivitis (GCP) worse than grade 1
    * Anterior uveitis or iritis (past or present)
    * Seborrheic eczema, Seborrheic conjunctivitis
    * History of corneal ulcers or fungal infections
    * Poor personal hygiene
  * Has a known history of corneal hypoesthesia (reduced corneal sensitivity)
  * Has aphakia, keratoconus or a highly irregular cornea.
  * Has Presbyopia or has dependence on spectacles for near work over the contact lenses.
  * Has undergone corneal refractive surgery.
  * Is participating in any other type of eye related clinical or research study.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2016-09; Primary Completion 2016-11 (Actual); Study Completion 2016-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Velázquez Guerrero, MSc., FIACLE, Principal Investigator — School of Optometry, National Autonomous University (UNAM)
Locations (1):
- Optometry Clinic, National Autonomous University, Mexico City, Mexico

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Filcon IV1 Toric Lens, Then Ocufilcon D Toric Lens: Participants are randomized to wear filcon IV1 toric lens, then ocufilcon D toric lens pair for 1 week each during the cross over study.
  filcon IV1: toric contact lens
  ocufilcon D: toric contact lens
- Ocufilcon D Toric Lens, Then Filcon IV1 Toric Lens: Participants are randomized to wear ocufilcon D toric lens, then filcon IV1 lens pair for 1 week each during the cross over study.
  filcon IV1: toric contact lens
  ocufilcon D: toric contact lens
Period: First Intervention (1 Week)
Arm/Group | Filcon IV1 Toric Lens, Then Ocufilcon D Toric Lens | Ocufilcon D Toric Lens, Then Filcon IV1 Toric Lens
Started | 15 | 15
Completed | 15 | 15
Not Completed | 0 | 0
Period: Second Intervention (1 Week)
Arm/Group | Filcon IV1 Toric Lens, Then Ocufilcon D Toric Lens | Ocufilcon D Toric Lens, Then Filcon IV1 Toric Lens
Started | 15 | 15
Completed | 15 | 15
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: There was 1 protocol deviation. Therefore, of the 30 subjects who completed the study, data from one subject is not included in the analysis.
Groups:
- Overall Participants: Participants are randomized to wear filcon IV1 or ocufilcon D toric lens pair for 1 week during the cross over study.
  filcon IV1: toric contact lens
  ocufilcon D: toric contact lens
Arm/Group | Overall Participants
Number analyzed (Participants) | 29
Age, Continuous [Mean (Standard Deviation); unit: years] | 27.7 (5.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21
  Male | 8

OUTCOME MEASURES:

1. Primary Outcome: Overall Fit Acceptance
Description: Investigator's preference for lens fit acceptance for habitual lenses assessed at baseline and filcon IV1 and ocufilcon D toric lenses assessed at baseline and 1 week. Scale 0-4, 0=should not be worn, 1=borderline but unacceptable, 2= minimally acceptable, early review, 3=not perfect but OK to dispense, 4=perfect
Time Frame: Baseline and 1 week
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Habitual Lens (Baseline): Habitual data was assessed at baseline.
- Filcon IV1 Toric Lens (Baseline); Filcon IV1 Toric Lens (1 Week): Participants are randomized to wear filcon IV1 toric lens pair for 1 week during the cross over study.
  filcon IV1: toric contact lens
- Ocufilcon D Toric Lens (Baseline); Ocufilcon D Toric Lens (1 Week): Participants are randomized to wear ocufilcon D toric lens pair for 1 week during the cross over study.
  ocufilcon D: toric contact lens
Arm/Group | Habitual Lens (Baseline) | Filcon IV1 Toric Lens (Baseline) | Ocufilcon D Toric Lens (Baseline) | Filcon IV1 Toric Lens (1 Week) | Ocufilcon D Toric Lens (1 Week)
Number analyzed (Participants) | 29 | 29 | 29 | 29 | 29
units on a scale | 3.8 (0.5) | 3.5 (0.5) | 3.7 (0.5) | 3.8 (0.4) | 3.7 (0.5)

2. Primary Outcome: Lens Centration
Description: Lens centration for habitual lenses assessed at baseline and filcon IV1 and ocufilcon D toric lenses assessed at baseline and 1 week. (Centered - optimal, decentered slightly, or substantially decentered).
Time Frame: Baseline and 1 week
Measure: Number; unit: percentage of participants
Groups:
- Optimal Centration; Decentered Slightly; Substantially Decentered: Lens centration
Arm/Group | Optimal Centration | Decentered Slightly | Substantially Decentered
Number analyzed (Participants) | 29 | 29 | 29
percentage of participants
  Habitual toric lens | 100 | 0 | 0
  Baseline - filcon IV1 toric | 100 | 0 | 0
  Baseline - ocufilcon D toric | 100 | 0 | 0
  1 week - filcon IV1 toric | 100 | 0 | 0
  1 week - ocufilcon D toric | 100 | 0 | 0

3. Primary Outcome: Post-blink Movement
Description: Post-blink movement for habitual lenses assessed at baseline and filcon IV1 and ocufilcon D toric lenses assessed at baseline and 1 week. Scale 0-4, 0=insufficient, 1=minimal, but acceptable movement, 2=optimal movement, 3=moderate, but acceptable movement, 4=excessive, unacceptable movement.
Time Frame: Baseline and 1 week
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Habitual Lens (Baseline): Habitual lens assessed at baseline.
Arm/Group | Habitual Lens (Baseline) | Filcon IV1 Toric Lens (Baseline) | Ocufilcon D Toric Lens (Baseline) | Filcon IV1 Toric Lens (1 Week) | Ocufilcon D Toric Lens (1 Week)
Number analyzed (Participants) | 29 | 29 | 29 | 29 | 29
units on a scale | 1.97 (0.5) | 2.1 (0.3) | 2.1 (0.4) | 2.0 (0.3) | 2.2 (0.4)

4. Primary Outcome: Overall Stability
Description: Overall lens stability for habitual lenses assessed at baseline and filcon IV1 and ocufilcon D toric lenses assessed at baseline and 1 week. Scale 0-4, 0=very poor stability, 4=excellent stability.
Time Frame: Baseline and 1 week
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Habitual Toric Lens: Habitual data was assessed at baseline.
- Filcon IV1 Toric Lens (Baseline): Data collected at baseline for filcon IV1 toric lens.
- Ocufilcon D Toric Lens (Baseline): Data collected at baseline for ocufilcon D toric lens.
- Filcon IV1 Toric Lens (1 Week): Data collected at 1 week for filcon IV1 toric lens.
- Ocufilcon D Toric Lens (1 Week): Data collected at 1 week for ocufilcon D toric lens.
Arm/Group | Habitual Toric Lens | Filcon IV1 Toric Lens (Baseline) | Ocufilcon D Toric Lens (Baseline) | Filcon IV1 Toric Lens (1 Week) | Ocufilcon D Toric Lens (1 Week)
Number analyzed (Participants) | 29 | 29 | 29 | 29 | 29
units on a scale | 3.8 (0.5) | 3.6 (0.5) | 3.8 (0.4) | 3.7 (0.5) | 3.7 (0.6)

5. Primary Outcome: Corneal Coverage
Description: Corneal coverage for habitual lenses assessed at baseline and filcon IV1 and ocufilcon D toric lenses assessed at baseline and 1 week. (yes=full corneal coverage or no=not full coverage)
Time Frame: Baseline and 1 week
Measure: Number; unit: participants
Groups:
- Filcon IV1 Toric Lens: Participants are randomized to wear filcon IV1 toric lens pair for 1 week during the cross over study.
  filcon IV1: toric contact lens
- Ocufilcon D Toric Lens: Participants are randomized to wear ocufilcon D toric lens pair for 1 week during the cross over study.
  ocufilcon D: toric contact lens
Arm/Group | Filcon IV1 Toric Lens | Ocufilcon D Toric Lens
Number analyzed (Participants) | 29 | 29
participants
  Habitual toric lens - Yes | 29 | 29
  Habitual toric lens - No | 0 | 0
  Baseline - Yes | 29 | 29
  Baseline - No | 0 | 0
  1 week - Yes | 29 | 29
  1 week - No | 0 | 0

6. Primary Outcome: Lens Orientation in Primary Position of Gaze
Description: Lens rotation for habitual toric lens assessed at baseline and filcon IV1 and ocufilcon D toric lenses assessed at baseline and 1 week with slit lamp by measuring within 10 degrees of the axis mark on the lens relative to the desired 6' o'clock position while the subject looked straight ahead.
Time Frame: Baseline and 1 week
Measure: Number; unit: percentage of participants
Groups:
- Habitual Toric Lens: Habitual data was gathered at baseline.
Arm/Group | Habitual Toric Lens | Filcon IV1 Toric Lens (Baseline) | Ocufilcon D Toric Lens (Baseline) | Filcon IV1 Toric Lens (1 Week) | Ocufilcon D Toric Lens (1 Week)
Number analyzed (Participants) | 29 | 29 | 29 | 29 | 29
percentage of participants
  0 degrees | 62 | 72 | 76 | 79 | 79
  <=5 degrees | 35 | 21 | 21 | 7 | 14
  <=10 degrees | 3 | 7 | 3 | 14 | 7

7. Primary Outcome: Rotational Recovery in Degrees After 60 Seconds
Description: Rotational recovery measured in degrees after 60 seconds for habitual toric lens assessed at baseline and filcon IV1 and ocufilcon D toric lenses assessed at baseline and at 1 week by slit lamp.
Time Frame: Baseline and 1 week
Measure: Mean (Standard Deviation); unit: degrees
Arm/Group | Habitual Toric Lens | Filcon IV1 Toric Lens (Baseline) | Ocufilcon D Toric Lens (Baseline) | Filcon IV1 Toric Lens (1 Week) | Ocufilcon D Toric Lens (1 Week)
Number analyzed (Participants) | 29 | 29 | 29 | 29 | 29
degrees | 4.1 (6.7) | 5.0 (7.1) | 3.3 (4.7) | 2.2 (4.1) | 3.8 (8.5)

ADVERSE EVENTS:
Arm/Group | Filcon IV1 Toric Lens | Ocufilcon D Toric Lens
All-Cause Mortality (participants affected / at risk) | 0/30 | 0/30
Serious Adverse Events (participants affected / at risk) | 0/30 | 0/30
Other Adverse Events (participants affected / at risk) | 0/30 | 0/30

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other